CLINICAL TRIAL: NCT05611671
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of 3 Active Dose Regimens of MORF-057 in Adults With Moderately to Severely Active Ulcerative Colitis (EMERALD-2)
Brief Title: A Study to Evaluate MORF-057 in Adults With Moderately to Severely Active UC
Acronym: EMERALD-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Therapeutic, Inc. (A Wholly Owned Subsidiary of Eli Lilly and Company) (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27398; J6E-MC-KWAD (Other: Eli Lilly and Company); MORF-057-202 (Other: Morphic Therapeutic, Inc); 2022-500953-17-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative
Keywords: Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD); a4b7; Moderate-to-severe; Integrin; EMERALD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MORF-057 200 mg BID (Experimental): Participants received a 200 milligram (mg) oral dose of MORF-057 twice daily (BID) for 12 weeks.
  Interventions: Drug: MORF-057
- MORF-057 100 mg BID (Experimental): Participants received a 100 mg oral dose of MORF-057 twice daily for 12 weeks.
  Interventions: Drug: MORF-057
- MORF-057 100 mg QD-M (Experimental): Participants received a 100 mg oral dose of MORF-057 once daily in the morning (QD-M) for 12 weeks.
  Interventions: Drug: MORF-057
- Placebo (Placebo Comparator): Participants received an oral dose of matching placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MORF-057 — MORF-057 is a small molecule that is designed to selectively inhibit integrin α4β7 and is administered orally.
  Other Names: LY4268989
  Arms: MORF-057 100 mg BID; MORF-057 100 mg QD-M; MORF-057 200 mg BID
Drug: Placebo — Matching placebo (identical appearance to MORF-057) administered orally.
  Arms: Placebo

SUMMARY:
This is a Phase 2b randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of three active dose regimens of MORF-057 in adult patients with moderately to severely active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
This is a Phase 2b randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of three active dose regimens of MORF-057 plus a placebo regimen in study participants with moderately to severely active UC. After completion of the 12-week Induction Period, participants may be switched to a different active MORF-057 regimen during the Maintenance Period. Those randomized into the placebo group in the Induction Period will be switched to receive an active MORF-057 regimen during the Maintenance Period.

ELIGIBILITY:
Inclusion Criteria:

* Has signs/symptoms of moderate to severe UC for at least 3 months prior to Screening
* Has evidence of UC extending at least 15 cm from the anal verge
* Demonstrated an inadequate response, loss of response, or intolerance to at least one of the following treatments: Oral aminosalicylates (e.g., mesalamine, sulfasalazine, olsalazine, or balsalazide), corticosteroids, immunosuppressants (e.g., azathioprine, 6-mercaptopurine, or methotrexate), advanced therapies for UC (e.g., biologic agents, Janus kinase [JAK] antagonists, or sphingosine-1-phosphate [S1P] receptor agonists)
* Subject has no prior exposure to approved or investigational anti-integrin therapies
* Agrees to abide by the study guidelines and requirements
* Capable of giving signed informed consent

Exclusion Criteria:

* Diagnosed with indeterminate colitis, microscopic colitis, ischemic colitis, radiation colitis, or Crohn's disease or has clinical findings suggestive of Crohn's disease
* Has positive findings on a subjective neurological screening questionnaire
* Has a concurrent, clinically significant, serious, unstable comorbidity
* Previous treatment with vedolizumab or other licensed or investigational integrin inhibitors
* Participation in any other interventional study or received any investigational therapy within 30 days
* Previous exposure to MORF-057 and/or a known hypersensitivity to drugs with a similar mechanism to MORF-057
* Unable to attend study visits or comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (8):
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Gastro Care Institute, Lancaster, California
  - TLC Clinical Research Inc., Los Angeles, California
  - Innova Clinical Trials, Coral Gables, Florida
  - Eminat, LLC - Miramar, Miramar, Florida
  - Robert Wood Johnson University Medical School, New Brunswick, New Jersey
  - Great Lakes Gastroenterology, Mentor, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Australia (5):
  - Blacktown Hospital, Blacktown
  - Concord Repatriation General Hospital, Concord
  - Royal Brisbane and Women's Hospital, Herston
  - Fiona Stanley Hospital, Murdoch
  - Mater Adult Hospital Brisbane, South Brisbane
- Austria (3):
  - Order Hospital Linz Ltd. - Hospital of Sisters of Mercy, Linz
  - Salzburg Regional Hospital, Salzburg
  - Medical University of Vienna, Vienna
- Bulgaria (4):
  - Medical Center "Rusemed" EOOD, Rousse
  - University Multiprofile Hospital for Active Treatment "ACIBADEM City Clinic", Sofia
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, Sofia
  - Second Multiprofile Hospital for Active Treatment - Sofia, Sofia
- Czechia (2):
  - PreventaMed, s.r.o., Olomouc
  - Clinoxus s.r.o., Outpatient Clinic Budejovicka, Prague
- Estonia (5):
  - LV Venter OU, Pärnu
  - OU Innomedica, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - University of Tartu, Tartu
- Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice, France
- Georgia (6):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
  - Curatio, Jsc, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - Medical Center "CITO" Ltd., Tbilisi
  - LTD The First Medical Center, Tbilisi
- Germany (4):
  - Charite - University Hospital Berlin, Berlin
  - Krankenhaus Waldfriede, Berlin
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital Ulm, Ulm
- Hungary (6):
  - Semmelweis Medical University, Budapest
  - Semmelweis University, Department of Internal Medicine and Haematology, Division of Internal Medicine and Gastroenterology, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
  - Fejer County St. Gyorgy University Teaching Hospital, Székesfehérvár
  - Javorszky Odon Korhaz, Vác
- India (10):
  - Fortis Memorial Research Institute(FMRI), Gūrgaon
  - Gleneagles Hospital, Hyderabad
  - Sawai Man Singh Medical College Hospital (SMS Hospital), Jaipur
  - S R Kalla Memorial Gastro and General Hospital, Jaipur
  - Dayanand Medical College and Hospital, Ludhiana
  - All India Institute of Medical Sciences, New Delhi
  - Fortis Hospital, Noida
  - Yashoda Hospital, Secunderabad
  - SIDS Hospital and Research Centre, Surat
  - Government Medical College, Thiruvananthapuram
- Israel (2):
  - Shaare Zedek Medical Center, Digestive Diseases Institute, Jerusalem
  - Kaplan Medical Center, Institute of Gastroenterology and Liver Diseases, Rehovot
- Italy (5):
  - Ospedale Luigi Sacco, Milan
  - Hospital of Padova, Padua
  - IRCCS Istituto Clinico Humanitas- Centro Malattie Infiammatorie Intestinali, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - IRCCS Ospedale San Raffaele, Segrate
- Latvia (3):
  - Liepaja Regional Hospital, Liepāja
  - Digestive Diseases Center "Gastro", Riga
  - Pauls Stradins Clinical Univeristy Hospital, Riga
- Lithuania (2):
  - Republican Panevezys Hospital, Panevezys
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (18):
  - CLINSANTE Clinical Research Centre Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - St. John Paul 2nd Municipal Hospital in Elblag, Elblag
  - "Vita Longa" Non-Public Healthcare Facility, Limited Liability Company, Katowice
  - Krakow Medical Center, Krakow
  - IP Clinic, Lodz
  - University Teaching Hospital No. 4 in Lublin, Lublin
  - ETG Lublin, Lublin
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - EMC Medical Institute Joint Stock Company, "Certus" Private Healthcare Facility Hospital No. 1, Poznan
  - Twoja Przychodnia Pcm, Poznan
  - Endoscopy Limited Liability Company, Sopot
  - New health-CK, Kieltucki and partners g.p., Staszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - H-T. Medical Center, Tychy
  - Centrum Medyczne Reuma Park, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - EMC Medical Institute Joint Stock Company, EuroMediCare Specialist Outpatient Clinics in Wroclaw, Wroclaw
  - ETG Zamość, Zamość
- Romania (2):
  - Colentina Clinical Hospital, Bucharest
  - Center of Diagnosis and Treatment Provita, Bucharest
- Serbia (3):
  - Zvezdara University Medical Center, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (3):
  - Cliniq s.r.o., Bratislava
  - ENDOMED s.r.o., Košice
  - Gastro LM s.r.o., Prešov
- South Korea (3):
  - Dong-A University Hospital, Busan
  - Yeungnam Univeristy Medical Center, Daegu
  - Kyung Hee University Hospital, Seoul
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chia-Yi Christian Hospital, Chiayi City
  - Tri-Service General Hospital, Neihu Taipei
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MORF-057 200 mg BID | MORF-057 100 mg BID | MORF-057 100 mg QD-M | Placebo
Started | 69 | 71 | 70 | 70
Safety Analysis Population (All participants who received at least one dose of the study drug. Participants were analyzed according to the treatment they actually received.) | 70 (One participant randomized to the placebo group inadvertently received 200 mg of MORF-057 and was therefore included in 'MORF-057 200 mg BID' arm for safety analyses.) | 71 | 70 | 69
Completed (Participants who completed the 12-week treatment were considered as 'completed.') | 65 | 68 | 67 | 65
Not Completed | 4 | 3 | 3 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- MORF-057 200 mg BID: Participants received a 200 mg oral dose of MORF-057 twice daily for 12 weeks.
- MORF-057 100 mg QD-M: Participants received a 100 mg oral dose of MORF-057 once daily in the morning for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | MORF-057 200 mg BID | MORF-057 100 mg BID | MORF-057 100 mg QD-M | Placebo | Total
Number analyzed (Participants) | 69 | 71 | 70 | 70 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (17.14) | 41.8 (14.35) | 38.9 (13.57) | 39.1 (13) | 40.2 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 31 | 34 | 125
  Male | 41 | 39 | 39 | 36 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 2 | 6
  Not Hispanic or Latino | 66 | 70 | 69 | 68 | 273
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 11 | 13 | 13 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 53 | 60 | 57 | 57 | 227
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission as Determined Using the Modified Mayo Clinic Score (mMCS)
Description: * The mMCS is a scoring system for assessment of ulcerative colitis activity and is a composite of Endoscopic subscore (range: 0=Normal or inactive disease to 3=Severe disease (spontaneous bleeding, ulceration)), Stool Frequency subscore (range: 0=Normal number of stools to 3=5 or more stools more than normal), and Rectal Bleeding subscore (range: 0=No blood seen to 3=Blood alone passed). The mMCS total score ranges from 0 to 9, with higher scores indicating more severe disease.
  * Clinical remission per mMCS is defined as rectal bleeding subscore of 0; a stool frequency subscore of < or =1; and an endoscopy subscore of < or =1 without friability.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | MORF-057 200 mg BID | MORF-057 100 mg BID | MORF-057 100 mg QD-M | Placebo
Number analyzed (Participants) | 69 | 71 | 70 | 70
percentage of participants | 31.9 | 23.9 | 17.1 | 24.3
Statistical Analysis 1: Comparison: MORF-057 200 mg BID vs Placebo; Test type: Other; Risk Difference (RD) = 6.71, 95% CI 2-sided [-7.76 to 21.18]
Statistical Analysis 2: Comparison: MORF-057 100 mg BID vs Placebo; Test type: Other; Risk Difference (RD) = -0.41, 95% CI 2-sided [-13.99 to 13.17]
Statistical Analysis 3: Comparison: MORF-057 100 mg QD-M vs Placebo; Test type: Other; Risk Difference (RD) = -6.93, 95% CI 2-sided [-19.74 to 5.88]

2. Secondary Outcome: Percentage of Participants in Clinical Response as Determined Using the Modified Mayo Clinic Score (mMCS)
Description: * The mMCS is a scoring system for assessment of ulcerative colitis activity and is a composite of Endoscopic subscore (range: 0=Normal or inactive disease to 3=Severe disease (spontaneous bleeding, ulceration)), Stool Frequency subscore (range: 0=Normal number of stools to 3=5 or more stools more than normal), and Rectal Bleeding subscore (range: 0=No blood seen to 3=Blood alone passed). The mMCS total score ranges from 0 to 9, with higher scores indicating more severe disease.
  * Clinical response per mMCS is defined as decrease from baseline in the mMCS score > or =2 points and > or =30% from baseline, plus a decrease in rectal bleeding subscore > or =1 or an absolute rectal bleeding subscore < or =1.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | MORF-057 200 mg BID | MORF-057 100 mg BID | MORF-057 100 mg QD-M | Placebo
Number analyzed (Participants) | 69 | 71 | 70 | 70
percentage of participants | 62.3 | 53.5 | 57.1 | 54.3
Statistical Analysis 1: Comparison: MORF-057 200 mg BID vs Placebo; Test type: Other; Risk Difference (RD) = 7.05, 95% CI 2-sided [-8.77 to 22.86]
Statistical Analysis 2: Comparison: MORF-057 100 mg BID vs Placebo; Test type: Other; Risk Difference (RD) = -0.93, 95% CI 2-sided [-16.74 to 14.88]
Statistical Analysis 3: Comparison: MORF-057 100 mg QD-M vs Placebo; Test type: Other; Risk Difference (RD) = 3.07, 95% CI 2-sided [-12.78 to 18.92]

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: All participants from the safety analysis population set.
Arm/Group | MORF-057 200 mg BID | MORF-057 100 mg BID | MORF-057 100 mg QD-M | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/70 | 3/71 | 0/70 | 1/69
Other Adverse Events (participants affected / at risk) | 9/70 | 8/71 | 5/70 | 10/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORF-057 200 mg BID (N=70) | MORF-057 100 mg BID (N=71) | MORF-057 100 mg QD-M (N=70) | Placebo (N=69)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORF-057 200 mg BID (N=70) | MORF-057 100 mg BID (N=71) | MORF-057 100 mg QD-M (N=70) | Placebo (N=69)
Headache (Nervous system disorders) | 5 | 4 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 4
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05611671/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT05611671/SAP_001.pdf